CLINICAL TRIAL: NCT00558597
Title: Proteomics Analysis for Recognition of Acute Cellular Rejection After Lung Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Hannover Medical School, Medical School
Other Study IDs: 154
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2008-09

CONDITIONS: Rejection; Lung Transplantation
Keywords: Proteomics; Lung Transplantation
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — BAL (broncho alveolar lavage) urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 30 patients with stable graft function
- 2: 30 patients with acute rejection after lung transplantation

SUMMARY:
In patients with acute rejection after lung transplantation the peptide profile in broncho-alveolar lavage (BAL) and urine should be compared in order to identify a paradigm that allows an non-invasive rejection therapy.

DETAILED DESCRIPTION:
Goal of the study is the establishment of biomarkers for early diagnosis of acute rejection, followed by a late validation of the paradigm with prospectively collected samples, which will be examined blinded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable graft function
* Patients with acute rejection

Exclusion Criteria:

* Acute infection
* BOS

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients after lung transplantation
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-03; Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Gottlieb, Dr. med., Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany